CLINICAL TRIAL: NCT06542328
Title: Pre-market Verification of Portable X Ray Machines for Lung Diseases and Orthopedic Limb
Brief Title: Pre-market Verification of Portable X Ray Machines for Lung Diseases and Orthopedic Limb Lesions
Status: Completed | Type: Observational
Sponsor: Energy Resources International Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 110A-305
Record Dates: First submitted 2024-07-31; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: X-rays; Effects; Chest--Diseases; Orthopedic Disorder
Keywords: Portable X ray machine; Extremities; Telemedicie
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pulmonology
  Interventions: Device: ERI CVX-air portable X-ray system; Device: Samsung GM85 (K180543) or MobileDaRt Evolution (K080701)
- Orthopaedic
  Interventions: Device: ERI CVX-air portable X-ray system; Device: Samsung GC85A (K160997) or Fujifilm FDR Smart X (K212956)

INTERVENTIONS:
Device: ERI CVX-air portable X-ray system — investigational device
Device: Samsung GM85 (K180543) or MobileDaRt Evolution (K080701) — The commercially available comparator equipment used for pulmonology.
  Groups: Pulmonology
Device: Samsung GC85A (K160997) or Fujifilm FDR Smart X (K212956) — The commercially available comparator equipment used for Orthopaedic.
  Groups: Orthopaedic

SUMMARY:
The clinical trial is to evaluate a portable X ray machine (model name: CVXair) for chest and extremities diagnosis, the performance of machine is comparing to the commercial stationary and portable machine both in biological structure way and disease diagnosis way by the image generated.

Currently sold X ray machines in market for hospital are stationary or big size portable, it is not easy for carrying to use and occupied a large space for installation and storage, beside that, CVXair is a small and light machine within 3.2KG and has extremely low dosage. It is the reason we expect to use CVXair as a convenient X ray machine with low radiation dosage for X ray image diagnosis clinically.

This trial has an expected trial period in two years, the accepted patients are limited to thoracic and orthopedics patients no matter out hospital or in hospital. The accepted patients upper limitation number is 123 respectively. The selected patient will be taken X ray shot in same area and position both by CVXair and market sold machine, the images then will be interpreted by 2 qualified radiologist in different biological structure and specified diseases. Then the process will be given by a suitable test score.

The test result will be calculated by defined index for comparing with the market sold X ray machines, and finally we will base on the result to state the machine is equivalent or not by the market sold X ray machines.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lung diseases and orthopedic limb lesions.
* Aged 20 years or older.
* After informed consent, sign the subject consent form.

Exclusion Criteria:

* Patients under the age of 20 years.
* Pregnant women (female subjects of childbearing potential, undergo pregnancy testing prior to irradiation to exclude the risk of pregnancy).
* Other individuals deemed unsuitable for inclusion in the clinical trial upon physician assessment.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects suspected of having pulmonary diseases or orthopedic limb disorders.
Sampling Method: Non-Probability Sample
Enrollment: 228 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-06-23 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Comparing the investigational device with the control device using Two Parellel-Sample Mean Test for Non-inferiority, the average scores of image quality at 5 anatomical sites. | Only images captured with the trial device and control device within a range of -1 day, 0 day, and 1 day from each other were selected for analysis.
  The average scores (Likert scale，1-4) for image quality at 5 anatomical sites/items generated by the investigational equipment for producing radiographic images of the thorax and limbs in human anatomy, compared to the commercial equipment, were evaluated based on the criteria defined in the study by Cheng Ting Lin et al. (Lin et al., 2020). These scores were assessed for diagnostic utility and level of defects.

CONTACTS AND LOCATIONS:
Locations (1):
- Changhua Christian Hospital, Changhua, Changhua County, Taiwan